CLINICAL TRIAL: NCT05896020
Title: Open, Multicenter Phase II Clinical Study of SHR-A1811 for Injection in the Treatment of Gynaecological Malignancies
Brief Title: A Study of SHR-A1811 in Subjects With Gynaecologic Oncology
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-209
Record Dates: First submitted 2023-05-28; First posted 2023-06-09 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Gynaecological Malignancies

STUDY DESIGN:
Intervention Model Description: Single arm study of SHR-A1811
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group with SHR-A1811 (Experimental)
  Interventions: Drug: SHR- A1811

INTERVENTIONS:
Drug: SHR- A1811 — Subjects with gynaecological malignancies

SUMMARY:
This is an open-label, two-part study to evaluate the safety and efficacy of SHR-A1811 for injection in subjects with a gynaecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and signed the ICF.
2. Measurable disease, as defined by RECIST v1.1.
3. The Eastern Cancer Cooperative Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 12 weeks.
5. Subjects with advanced cervical cancer, recurrent ovarian cancer and endometrial cancer.

Exclusion Criteria:

1. Symptomatic, untreated or active central nervous system metastases.
2. Previously received antibo-conjugated drugs with the following characteristics: topoisomerase I inhibition in the composition Preparations, such as Enhertu (DS-8201a), U3-1402, etc..
3. Have uncontrolled or severe cardiovascular disease.
4. With any active autoimmune disease or history of autoimmune disease.
5. Patients with active hepatitis B or hepatitis C.
6. Severe infections within 28 days prior to initiation of study treatment.
7. Active tuberculosis within one year prior to initiation of study treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | 12 months
Objective response rate (ORR) | 12 months
Disease control rate (DCR) | 12 months
Duration of response (DOR) | 12 months
Overall survival (OS) | 12 months
Incidence and severity of adverse events (AEs) | From Day 1 to 90 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided